CLINICAL TRIAL: NCT01761968
Title: Long-term Study Evaluating the Effect of Givinostat in Patients With JAK2V617F Positive Chronic Myeloproliferative Neoplasms
Brief Title: Long-term Study Evaluating the Effect of Givinostat in Patients With Chronic Myeloproliferative Neoplasms
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSC/11/2357/44; 2012-003499-37 (EudraCT Number)
Record Dates: First submitted 2012-12-18; First posted 2013-01-07 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Chronic Myeloproliferative Neoplasms
Keywords: chronic myeloproliferative neoplasms; Polycythemia Vera; Essential Thrombocythemia; Primary Myelofibrosis; Post-Polycythemia Vera Myelofibrosis; Post-Essential Thrombocythemia Myelofibrosis; Givinostat
MeSH Terms: conditions — Myeloproliferative Disorders; Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis | interventions — givinostat; givinostat hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- givinostat (Experimental): Patients will continue at their last tolerable dose and treatment schedule of givinostat monotherapy. Givinostat is a histone-deacetylases inhibitor. The product will be supplied as hard gelatine capsules for oral administration at the strength of 50 mg, 75 mg and/or 100 mg each.
  If patients previously received givinostat in combination with other drugs during a core protocol or a compassionate use program, they will be treated at their last tolerable dose of this combination.
  Interventions: Drug: givinostat

INTERVENTIONS:
Drug: givinostat — Patients will continue at their last tolerable dose and treatment schedule of givinostat monotherapy. Givinostat is a histone-deacetylases inhibitor. The product will be supplied as hard gelatine capsules for oral administration at the strength of 50 mg, 75 mg and/or 100 mg each.
  If patients previously received givinostat in combination with other drugs during a core protocol or a compassionate use program, they will be treated at their last tolerable dose of this combination.
  Other Names: givinostat (ITF2357)

SUMMARY:
This is a multicenter, open label, long-term study testing the long-term safety, tolerability and efficacy of givinostat in patients with Polycythemia Vera, Essential Thrombocythemia, primary Myelofibrosis, Post-Polycythemia Vera Myelofibrosis, Post-Essential Thrombocythemia Myelofibrosis following core protocols in chronic myeloproliferative neoplasms and/or patient-named compassionate use program (if regulated/allowed by the local regulations, e.g. for Italy D.M. 8/5/2003 "Uso terapeutico di medicinale sottoposto a sperimentazione clinica" published on G.U. n. 173 of 28 July 2003, and the following amendments). Patients will continue at their last tolerable dose and treatment schedule of givinostat monotherapy. If patients previously received givinostat in combination with other drugs during a core protocol or a compassionate use program (if regulated/allowed by the local regulations, e.g. for Italy D.M. 8/5/2003 "Uso terapeutico di medicinale sottoposto a sperimentazione clinica" published on G.U. n. 173 of 28 July 2003, and the following amendments), they will be treated at the last tolerable dose of the combination. Assessment of safety and efficacy will be performed at each quarterly visit and each visit will also include laboratory tests and ECG examination. During the visits the clinical benefit will be assessed by Investigator according to the revised European LeukemiaNet response criteria (for PV and ET) and EUMNET response criteria (for MF). The dose of Givinostat will be modified for protocol specified toxicities. The treatment may continue up to Marketing Authorization of givinostat, currently planned in the next 5 years (note: only for Germany, this long-term study is initially limited up to 2 years of treatment). Patients may discontinue study treatment at any time and remain on study therapy as long as they derive clinical benefit. Safety will be monitored at each visit throughout the entire duration of the study. In case the approved label will not cover the whole study population, givinostat will be provided by the Sponsor to those patients not fulfilling the criteria for the approved label of the drug that are still deriving benefit from givinostat at the time of its commercial availability.

DETAILED DESCRIPTION:
This is a multicenter, open label, long-term study testing the long-term safety, tolerability and efficacy of givinostat in patients with PV, ET, primary MF, Post-PV MF, Post-ET MF following core protocols in cMPN (i.e. Study DSC/07/2357/28, Study DSC/08/2357/38, Study DSC/12/2357/45 and/or all further core protocols in cMPN), and/or patient-named compassionate use program (if regulated/allowed by the local regulations, e.g. for Italy D.M. 8/5/2003 "Uso terapeutico di medicinale sottoposto a sperimentazione clinica" published on G.U. n. 173 of 28 July 2003, and the following amendments).

Eligible patients will have tolerated previous givinostat treatment and achieved a clinical benefit at the end of the core protocols; alternatively, eligible patients are participating in compassionate use program (if regulated/allowed by the local regulations, e.g. for Italy D.M. 8/5/2003 "Uso terapeutico di medicinale sottoposto a sperimentazione clinica" published on G.U. n. 173 of 28 July 2003, and the following amendments). In addition, patients must have tolerated previous givinostat treatment and achieved a clinical benefit at the end of core protocols or compassionate use program with givinostat, assessed by the Investigator according to the revised clinico-haematological ELN response criteria (for PV and ET) and EUMNET response criteria (for MF).

After providing informed written consent before undertaking any protocol-related procedure, an unique patient identification code (patient ID) will be assigned to each patient, will identify the patient throughout his/her participation in the study and can never be reused in case of premature drop-out.

Patients will continue at their last tolerable dose and treatment schedule of givinostat monotherapy. If patients previously received givinostat in combination with other drugs (e.g. hydroxyurea) during a core protocol or a compassionate use program , they will be treated at the last tolerable dose of the combination. In general, the dose of study drug may not be increased during this study. However, since the Maximum Tolerated Dose (MTD) of givinostat as chronic treatment has been recently identified and proven tolerable in Polycythenia Vera patients (i.e. 100 mg b.i.d.), selected patients may be eligible for escalation of their givinostat dose up to this level upon consultation with and written permission by Italfarmaco S.p.A. or its designee.

Assessment of safety and efficacy will be performed at each quarterly visit and each visit will also include laboratory tests and ECG examination. During the visits the clinical benefit will be assessed by Investigator according to the revised clinico-haematological ELN response criteria (for PV and ET) and EUMNET response criteria (for MF). Patients will be considered for continued treatment on the basis of their clinical response:

* if patients continue to derive clinical benefit from participating in the study, they will be allowed to continue study medication;
* if patients do not derive clinical benefit from participating in the study, they will discontinue study treatment.

For patients who previously participated in a compassionate use program with Givinostat the decision to continue treatment will be based on the assessment of continued clinical benefit derived from study therapy.

Of note, since this is a long-term study, at each quarterly visit the Investigator should include in his/her clinical evaluation the patient's benefit-risk assessment, taking into account both the clinical course of the patient in the Study until the visit time (i.e. the "clinical benefit", as above defined in this paragraph) and also any possible treatment option available at the time when the visit is performed.

The dose of givinostat will be modified for protocol specified toxicities. The treatment may continue up to Marketing Authorization of Givinostat, currently planned in the next 5 years (note: only for Germany, this long-term study is initially limited up to 2 years of treatment).

Patients may discontinue study treatment at any time and remain on study therapy as long as they derive clinical benefit. Safety will be monitored at each visit throughout the entire duration of the study. Treatment will be administered on an outpatient basis and patients will be followed regularly with physical and laboratory tests, as specified in the protocol; in case of hospitalization, the treatment will be continued or interrupted according to the Investigators' decision.

In case the approved label will not cover the whole study population, givinostat will be provided by the Sponsor to those patients not fulfilling the criteria for the approved label of the drug that are still deriving benefit from Givinostat at the time of its commercial availability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have completed givinostat treatment on at least one core study in chronic myeloproliferative neoplasms, or patients must be participating in a compassionate use program with givinostat AND Patients must have tolerated previous givinostat treatment and achieved a clinical benefit at the end of core protocols or compassionate use program with givinostat, assessed by the Investigator according to the revised clinico-haematological ELN response criteria (for PV and ET) and EUMNET response criteria (for MF);
2. Patients must be able to provide informed consent and be willing to sign an informed consent form;
3. Adult patients (age ≥ 18 years) of both genders with established diagnosis of chronic myeloproliferative neoplasms according to the revised WHO criteria;
4. Patients must have an Eastern Cooperative Oncology Group performance status < 3 at baseline;
5. Acceptable organ function within 7 days of initiating study drug;
6. Use of an effective means of contraception for women of childbearing potential and men with partners of childbearing potential;
7. Willingness and capability to comply with the requirements of the study.

Exclusion Criteria:

1. Pregnancy or nursing (lactating) women, where pregnancy is defined as the state of a female after conception, confirmed by a positive human Chorionic Gonadotropin (hCG) laboratory test (i.e. > 5 mIU/mL) and until the termination of gestation;
2. A clinically significant corrected QT interval prolongation at baseline;
3. Use of concomitant medications known to prolong the corrected QT interval;
4. Clinically significant cardiovascular disease including:

   * Uncontrolled hypertension, myocardial infarction, unstable angina at screening;
   * New York Heart Association Grade II or greater congestive heart failure;
   * History of any cardiac arrhythmia requiring medication (irrespective of its severity);
   * A history of additional risk factors for Torsade de Point;
5. Active virus infection including human HIV, HBV and HCV;
6. Platelets count < 100 x109/L within 14 days before enrolment (i.e. the receipt of the Patient ID);
7. Absolute neutrophil count < 1.2 x109/L within 14 days before enrolment (i.e. the receipt of the Patient ID);
8. Total serum bilirubin > 1.5 1.5 x ULN except in case of Gilbert's disease or pattern consistent with Gilbert's disease;
9. Serum Aspartate aminotransferase/Alanine aminotransferase (AST/ALT) > 3 times the upper normal limit;
10. Serum Cystatin C > 2 x ULN for two subsequent evaluations (i.e. if the value of serum Cystatin C is >2 x ULN, the test will be repeated once, and if the value is again > 2 x ULN, this becomes an exclusioncriterion);
11. Uncontrolled hypertriglyceridemia at baseline, i.e. triglycerides ˃ 1.5 x ULN in fasting state.
12. History and/or presence of other diseases, metabolic dysfunctions, physical examination findings, or clinical laboratory findings giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the patient at high risk from treatment complications or significantly alter the absorption of the study drug;
13. Any investigational drug other than givinostat within 28 days before enrolment. Notably, the use of such medications within 28 days or 6 half-lives - whichever is longer - prior to the first dose of study drugs (i.e. Day 1) and during the study through all the study conduct (including any safety follow-up [FU] visit) is prohibited;
14. Use of concomitant medications known to inhibit Pgp;
15. Patients with known hypersensitivity to the components of potential study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Long-term safety and efficacy | 3 months
  To obtain information on the long-term safety and tolerability of givinostat in patients with chronic myeloproliferative neoplasms following core protocols or compassionate use program:
  * Number of patients experiencing adverse events;
  * Type, incidence, and severity of treatment-related adverse events.
  To determine the long term efficacy of givinostat in patients with chronic myeloproliferative neoplasms following core protocols or compassionate use program:
  * For Polycythemia Vera and Essential Thrombocythemia, Complete response and partial response rate according to the revised clinico-haematological European LeukemiaNet response criteria;
  * For Myelofibrosis, complete response, major response, moderate response and minor response rate according to European Myelofibrosis Network response criteria.
  Note that these assessment will be repeated periodically (each 3 months) during the study. In fact, the treatment will continue up to Marketing Authorisation of givinostat.

OTHER OUTCOMES:
Clinical exploratory endpoint | 1 year
  To evaluate the effect of givinostat on each single response parameter according to the revised European LeukemiaNet (for Polycythemia Vera and Essential Thrombocythemia) and European European Myelofibrosis Network response criteria (for Myelofibrosis).
  Note that this assessment will be repeated periodically (each year) during the study. In fact, the treatment will continue up to Marketing Authorisation of givinostat.
Molecular exploratory endpoint | 1 year
  To evaluate the molecular response (i.e. reduction of the allele burden of the mutated Janus Kinase 2 in the position V617F).
  Note that this assessment will be repeated periodically (each year) during the study. In fact, the treatment will continue up to Marketing Authorisation of givinostat.
Biomolecular exploratory endpoint | 1 year
  To identify potential other markers predictive of clinical benefit of givinostat (e.g. potential pharmacodynamic markers).
  Note that this assessment will be repeated periodically (each year) during the study. In fact, the treatment will continue up to Marketing Authorisation of givinostat.
Progression Free Survival | 1 year
  To evaluate the disease parameters related to disease evolution
Thrombotic Rate | 1 year
  To evaluate thrombotic rate

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Rambaldi, MD, Principal Investigator — Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, Italy
Locations (15):
- Germany (2):
  - Charite Research Organization GmbH, Berlin
  - Universitaetsklinikum Freiburg, Innere Medizin I - Haematologie und Onkologie, Freiburg im Breisgau
- Italy (11):
  - Azienda Ospedaliero-Universitaria Policlinico Consorziale, Bari, Bari, BA
  - Istituto Tumori Giovanni Paolo II IRCCS Ospedale Oncologico di Bari, Bari, BA
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo, BG
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Florence, FI
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico UOS Oncoematologia anziano, Milan, MI
  - Azienda Unità Sanitaria Locale - Presidio Ospedaliero "Spirito Santo", Pescara, Pescara, PE
  - Fondazione I.R.C.C.S.-Policlinico San Matteo, Pavia, Pavia, PV
  - Azienda Ospedaliera "Bianchi-Melacrino-Morelli", Reggio Calabria, RC
  - Ospedale San Bortolo, Vicenza, Vicenza, VI
  - Azienda Ospedaliera Universitaria Università degli Studi "Federico II", Naple, Naples
  - Università "Campus Bio-Medico", Rome, Rome
- United Kingdom (2):
  - Belfast City Hospital, Belfast
  - Royal Cornwall Hospital, Truro